CLINICAL TRIAL: NCT02753972
Title: Mindful Eating and Living: A Controlled Study Investigating the Effects of Mindfulness on Weight Loss, Habits, Mood and Biological Markers of Inflammation and Metabolism in Obese Post-Menopausal Women
Brief Title: Mindful Eating and Living for Obese Women
Acronym: MEAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This research was completed before January 18, 2017, and does not meet the ACT requirement to register and report results per the guidance provided in "Clinical Trials Registration and Results Information Submission" dated 09/21/2016.
Sponsor: University of New Mexico (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Brian Shelley, Family Practice Physician, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HRRC#: 06-254
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindful Eating and Living (Experimental): The goal of the Mindful Eating and Living (MEAL) intervention was to apply mindfulness to apply mindfulness to eating behavior. The content for the MEAL sessions included group discussion, mindfulness meditation, and group eating exercises. The course, based on the work of Kristeller, Baer, & Quillian-Wolever (31), emphasized brief daily meditation and pairing meditation with eating, but was more streamlined in terms of didactic content and course length. Participants examined hunger and satiety cues, the qualities of foods they crave, and emotional and cognitive states associated with eating. Each session included an eating exercise with a variety of foods. The monthly refresher sessions included a brief meditation, a brief eating exercise, and group discussion. (The MEAL curriculum is available from the authors.)
  Interventions: Behavioral: Mindful Eating and Living
- Active Control (Active Comparator): The Active Control (CONT) group matched the MEAL group regarding schedule. The agenda for the CONT sessions involved giving each participant the opportunity to discuss issues such as food choices, activity levels, and caloric goals. The sessions began by having the participants check-in about their experiences with eating. Next, the clinical psychology graduate student led the participants in goal setting and finally there was a question and answer period when the registered dietician answered questions about food selection. The monthly refresher sessions had the same agenda as the initial weekly sessions.
  Interventions: Behavioral: Active Weight Loss Control

INTERVENTIONS:
Behavioral: Mindful Eating and Living — 8 week mindfulness skills intervention
  Arms: Mindful Eating and Living
Behavioral: Active Weight Loss Control — 8 week active weight loss control group
  Arms: Active Control

SUMMARY:
Background: Mindfulness-based interventions may be effective in reducing the stress that may increase both obesity and inflammation.

Purpose: The purpose of this study was to examine the effects of a mindful eating intervention on weight loss and health-related outcomes.

Methods: Thirty-six obese, postmenopausal women were randomized to a six-week Mindful Eating and Living (MEAL) intervention or an active control group (CONT) consisting of nutritional counseling, goal setting, and group support. Weight, body mass index (BMI), waist-hip ratio (WHR), binge eating, interleukin-6 (IL-6) and C-reactive protein (CRP) were assessed at baseline and four follow-up periods up to one year.

Results: Multilevel analyses showed that the MEAL group had reductions in weight, BMI, WHR, binge eating, IL-6, and CRP; the CONT group had reductions in weight, BMI, and binge eating. The reductions in binge eating, IL-6, and CRP were greater for the MEAL as compared with the CONT group.

Conclusions: This study suggests that a mindfulness-based eating intervention may promote weight loss and reduce a variety of health-related risk factors in post-menopausal women who are obese.

DETAILED DESCRIPTION:
Hypothesis A brief mindfulness-based educational program specifically designed for obese individuals will enable them to gain mastery over previously automatic eating and activity habits and will be associated with enhanced mood, decreased inflammation, improved metabolic markers and weight control.

Specific Aims

1. To determine if a mindfulness-based educational program for obese persons (BMI ≥30) seeking to gain more control over eating and lifestyle result in significant improvement in BMI compared to a control group.
2. To determine if a mindfulness-based educational program for obese persons seeking to gain more control over eating and lifestyle result in significant improvements in insulin resistance and other metabolic and physiologic parameters.

   EXPERIMENTAL DESIGN AND METHODS

   The final design of this study will be influenced by the results of the pilot study entitled Mindful Eating and Living I (MEAL I), which is currently underway. After completing the analysis of data from MEAL I, 50 post-menopausal women between the ages of 55 and 70 with BMI ≥30 kg/m2 will be recruited and screened to allow for possible screen failures. The goal is to enroll a group of 40 participants (n=20 control, n=20 intervention).

   Randomization Study subjects will be randomized to treatment or control group and then further to an outpatient or inpatient admission subset. Randomization will be determined based on a randomization code devised by the University of New Mexico General Clinical Research Center (GCRC) statistician, and this randomization process will be administered by a GCRC staff person such that Drs. Sloan and Colleran, the investigators involved in the biological aspects of the study, will be blinded to the randomization.

   Enrolled subjects will be randomized as follows. Twenty will be randomized to the treatment group and 20 will be randomized to the control group. Those in the treatment group will receive counseling by the GCRC dietician as well as mindfulness training via the mindfulness curriculum developed during the MEAL 1 pilot study. Those in the control group will receive counseling by the GCRC dietician and monthly group check-in sessions. All subjects will have four GCRC visits to evaluate metabolic and physiologic parameters and to complete psychometric questionnaires.

   In-patient and Out-patient GCRC subsets Of the 40 enrolled subjects, 24 will be randomly assigned to a subset of patients who will be admitted for overnight stays in order to test insulin resistance parameters and to monitor nocturnal blood pressure. The remaining 16 subjects will have GCRC outpatient visits only. The rationale for an in-patient subset is logistical. Our protocol calls for patients to be admitted for baseline evaluation at a uniform time preceding the mindfulness intervention, and then at three later time points. All patients need to be evaluated as close to the same time as possible, as they are going through the intervention according to the same schedule. It is not logistically possible to admit 40 patients for overnight stays within a 10-14 day interval at four different time periods. Admitting a subset of 24 patients for overnight stay allows an adequate sample size to measure insulin resistance. The biological markers being measured require a larger sample size to show statistical significance, and this larger sample size can be achieved without inpatient stays.

   Screening Subjects will be screened in the outpatient GCRC. Screening procedures will include thyroid stimulating hormone and late night salivary cortisol to rule out secondary causes of obesity and a basic metabolic panel to rule out other untreated medical conditions. Other screening tests will include a history and physical, to ascertain ability to initiate an exercise program. As part of the physical exam, a mini mental status exam will be performed to screen for cognitive impairment that would preclude them from participating in the mindfulness training curriculum.

   Study Design All subjects will undergo an initial GCRC visit, which will be outpatient or inpatient based on their subset assignment. At this first visit, medical evaluation, psychometric questionnaire administration and laboratory evaluation will occur as detailed below. Because fasting is required for the lab draws, the outpatient subjects will then be given a snack or meal by the GCRC dietician. Subjects will then meet with the GCRC dietician for a one-hour counseling session on weight loss.

   Those subjects in the inpatient subset will not visit the out-patient GCRC. Instead, they will be admitted for an observed overnight fast followed by an oral glucose tolerance test and will also undergo frequent blood pressure monitoring. During this admission, the same information obtained from the out-patient subset of subjects will also be obtained, and just as with the out-patient subset, these subjects will have a one-hour counseling session with the GCRC dietician. These dietician sessions are modeled after standard of care and include education about the food pyramid, food choices, activity monitoring, food diary and determination of a caloric goal and weight goal.

   After the first GCRC visit, subjects randomized to the treatment group (n=20) will begin a 6-week two-hour course on mindful eating entitled Mindful Eating & Living (MEAL). MEAL is a mindfulness training program which is designed specifically for obese individuals. MEAL teaches skills which can lead to increased awareness of eating, emotions, and judgment. Also included is information about activity and nutrition. The goal of mindfulness training is to allow people to cultivate awareness of their behaviors and provide themselves with choices, resulting in less bingeing or overeating, as well as increased sense of control, improved mood, and eventually, reduced weight. MEAL is a 6-week curriculum, taught in weekly sessions of 2-hours each to a group of 20 people. Specific exercises include group discussion, mindfulness meditation, and group eating exercises. Participants use written materials and CD's at home on a daily basis. At the completion of the course, treatment subjects will then attend monthly refresher sessions.

   Subjects randomized to the control group will not undergo mindfulness training. In order to provide a socially supportive environment similar to that experienced by the treatment subjects, monthly check-in sessions will be conducted for the control subjects. At these sessions, subjects will be invited to check-in about their experiences with weight loss efforts including food choices, activity levels and caloric goals. The first check-in session will occur during week 1 of the treatment group's mindfulness course, the second during week 6 of the mindfulness course, after which monthly sessions will be held during the same weeks as the mindfulness refresher sessions.

   All subjects will undergo three additional outpatient or inpatient GCRC visits: #2) at the time of completion of the 6-week mindfulness training, #3) at the time four weeks after the final refresher course and #4) at the time three months after the final refresher course. The subjects of both the control and treatment groups will undergo GCRC visits during the same two-week period. All measures obtained at the first visit will be repeated. All subjects will have one-hour meetings with the GCRC dietician for weight loss counseling at each visit. The purpose of these GCRC visits or admissions will be to determine the immediate effects, short-term effects and long-term effects of the intervention on metabolic, inflammatory, and adipocytokine parameters. Out-patient subjects will be given their questionnaires in advance so they can complete them at their convenience and decrease the time required for their out-patient visits.

   Demographics data will be obtained at baseline. The following data will be obtained at baseline and at the three subsequent GCRC inpatient or outpatient visits: medical history, medication profile, smoking status, vital signs, body mass index (BMI), waist/hip measurements, bioelectrical impedance analysis (BIA), dual-energy X-ray absorptiometry (BXA), Neuroticism (Benet-Martinez), Perceived Stress (Cohen), Psychological Well-being Scale (Ryff), Resilience (Connor), Trait Meta-Mood Scale (Salovey), Physical Symptoms (Moos), Positive and Negative Affect (Watson), Spirituality and Religion (Fetzer), Kentucky Inventory of Mindfulness Skills (Baer), Freiburg Mindfulness Inventory (FMI; Buchheld), Beck Depression Inventory (Beck), Beck Anxiety Inventory (Beck), Binge Eating Scale (Gormally), Eating Inventory (Stunkard). At the post-mindfulness training visits, a meditation log will be collected from the treatment group subjects (attached). Psychometric data will be analyzed in Logan Hall of UNM's main campus.

   BIOLOGICAL MEASURES

   The following biological data will be obtained from blood samples, totaling approximately two teaspoons from each patient. Each of the following measures will be obtained at baseline and then at three additional time points as previously described.

   Insulin Sensitivity:

   Obesity is highly correlated with insulin resistance. Similarly, weight loss improves insulin sensitivity.30 Fasting glucose and insulin concentrations can be used to estimate the severity of insulin resistance (the HOMA model).41 A second validated measure of insulin resistance is the insulin resistance index (IRIp) which uses the formula: peak of blood glucose after oral glucose load x plasma insulin level/10.56 For this study subjects will fast for 12 hours glucose and insulin will be Measured at baseline (HOMA) and at 120 minutes (IRIp). We anticipate that MEAL will lead to significant improvements in insulin sensitivity. Literature review reveals that identifying a 40% decrease in HOMA-IR, given a large effect size, requires a sample size of 24, with 12 in each group.33,34 To see a 20% decrease in IRIp, given its medium to large effect size, requires a sample size of greater than 24.56 Nevertheless, identifying trends in IRIp is valuable. Furthermore, it is difficult to predict the change in insulin resistance we might see as a result of MEAL, as published studies involving drug and surgical interventions are poor comparisons.

   Fasting lipid profile:

   Along with insulin resistance, obesity is associated with a specific dyslipidemia including hypertriglyceridemia, low high-density lipoprotein (HDL) cholesterol and small dense and oxidized low-density lipoprotein (LDL) cholesterol.42-44 Weight reduction leads to significant improvements in hypertriglyceridemia.30 We anticipate that mindfulness will similarly improve lipid profiles. In order to see a statistically significant reduction in triglyceride levels of approximately 30%, given the medium to large effect sizes seen in the literature, requires a sample size of 40 with 20 in each group.33,34

   Adiponectin:

   Adiponectin is an adipose-derived protein that negatively correlates with increasing adiposity, insulin resistance, inflammatory mediators and cardiovascular disease. 31-33, 45 Recently, a significant increase in adiponectin levels was seen in obese women following gastric bypass surgery, resulting in improvements in insulin sensitivity.33 A thorough literature search has revealed that the effects of mindfulness practice on adipocytokine levels have not yet been investigated. The MEAL study hypothesizes that mindfulness practice will be associated with an increase in adiponectin related to predicted weight loss. While the MEAL intervention is different from the diet and surgical interventions currently cited in the literature, we predict that our sample size of 40 will be adequate to identify a statistically significant increase in adiponectin of approximately 50%, given the medium to large effect size seen in the literature.33,40

   Interleukin (IL)-6, tumor necrosis factor-alpha (TNF- α), highly sensitive CRP (C-reactive protein):

   CRP is a major marker of inflammation. Its production by the liver is stimulated by a network of adipocytokines including IL-6 and TNF- α.33, 35, 36 Type 2 diabetes has been shown to be preceded by a state of sub-clinical inflammation.35 Additionally, The European Prospective Investigation into Cancer and Nutrition (EPIC) Potsdam Study showed that increased levels of IL-6 independently predicted the risk of type 2 diabetes, and that a combined elevation of IL-6 and TNF-α was also associated with increased risk.35 Weight loss has been shown to induce a significant decrease in CRP and IL-6 and is associated with an improvement in insulin sensitivity.34 As well, a one-year multidisciplinary weight reduction program showed a decrease in IL-6 as well as TNF-α.37 MEAL thus proposes that mindfulness-associated weight reduction will be associated with a decrease in IL-6, TNF- α and high sensitive CRP, which will further be associated with improved insulin sensitivity as estimated by fasting insulin and fasting glucose.

   A linear correlation between IL-6 and age has been established with an increase of 0.016 pg/ml per year of life.47 This has not been found to be true for CRP. Previous studies show a 40-50% decrease in IL-6 and CRP with weight loss and display medium to large effect sizes.33,35 The effect size for TNF- α is much smaller.33,35 Thus, we predict that we will be able to identify a statistically significant decrease in IL-6 and CRP with a sample size of 40, while it will be unlikely that our TNF- α results will reach significance. Nevertheless, TNF- α is a central player in the adipocytokine cascade, and identifying trends in the relationships between TNF- α and the other markers remains a valuable endeavor. The normal increase of IL-6 with age will be accounted for in our analysis by entering age as a covariate.

   Plasminogen activator inhibitor type 1 (PAI-1):

   PAI-1 is an adipocytokine that negatively regulates fibrinolysis thus increasing thrombus formation. Its connection to cardiovascular disease, insulin resistance and type 2 diabetes has been previously established.38,39 Weight loss is associated with a decrease in PAI-1.29 Recently, the Health, Aging and Body Composition Study showed PAI-1 to be independently associated with incident diabetes, and this association did not vary by sex or race.40 We hypothesize that PAI-1 levels will decrease with mindfulness practice and will be associated with improved insulin sensitivity. To see a decrease of 30% in PAI-1 levels, given the medium to large effect sizes seen in the literature, requires a sample size of at least 40.40

   Cortisol States of glucocorticoid excess are known to be associated with insulin resistance and increased cardiovascular risk. Cortisol production has an adrenocorticotropic hormone (ACTH) dependent circadian rhythm with peak levels in the early morning and a nadir at night. ACTH and cortisol are secreted independent of circadian rhythm in response to physical and psychological stress.51 A previous study examining the transcendental meditation and cardiovascular risk revealed decreased cortisol levels.8 A study that has not yet been published by Waters et al hypothesizes that cortisol rhythmicity and response to meals is altered in obesity.57 We hypothesize that mindfulness training will result in decreased late night salivary cortisol levels and decreased serum cortisol levels in response to a glucose challenge.

   The following anthropometric and physiologic parameters will be obtained:

   Body Mass Index The Primary outcome will be a change in body mass index (BMI). Preliminary statistical analysis reveals that to show a statistically significant decrease in BMI of 1.25 points, given the large effect size, requires a sample size of 24 subjects, 12 in each group, to achieve 80% power with an alpha of 0.05. Our sample size of 40 is adequate to determine if there is a significant improvement in BMI. BMI will be measured and recorded at each study visit.

   Bioelectrical Impedance Analysis Bioelectrical impedance analysis (BIA) is a tool to measure total body fat mass.52 While our sample size is not adequate to measure significant changes in total body fat, previous experience has demonstrated that for publication in peer reviewed journals, multiple anthropometric measurements are beneficial even if they do not change significantly. As this test if fairly ease to perform and of no risk to subjects we propose to include it in our study design.

   Dual Energy X-ray Absorptiometry Dual energy x-ray absorptiometry (DEXA) is a method to measure body composition which has superior accuracy over other methods such as BIA or BMI.52,53 DEXA also has the capacity to measure fat in different compartments including central and peripheral. Given the small effect size seen in previous studies in measuring percent body fat, our sample size may be only adequate enough to show a trend in changes in this measure. Of equal importance, however, is change in body fat distribution. Abdominal adiposity is known to be a strong predictor of Insulin resistance.54 We therefore hypothesize that mindfulness training will result in a decreased amount of abdominal compared to peripheral adiposity.

   Waist to Hip Ratio Numerous studies have demonstrated that increases waist hip ratios represent a significant risk for metabolic syndrome and cardiovascular disease (CVD), independent of BMI. While our sample size is not adequate to measure significant changes in total body fat, previous experience has demonstrated that for publication in peer reviewed journals, multiple anthropometric measurements are beneficial even if they do not change significantly. As this test if fairly ease to perform and of no risk to subjects we propose to include it in our study design.

   Nocturnal blood pressure dip:

   Most individuals exhibit circadian variation in blood pressure with decreased night-time blood pressure.47 Previous studies have shown that in patients with or without hypertension, a diminished nocturnal decline in blood pressure is a risk for cardiovascular mortality and is associated with elevated levels of inflammatory markers including PAI-1.48, 49 To determine the effect of mindfulness training on nocturnal dip in blood pressure, we will admit a subset of patients for overnight stays and will monitor their blood pressure via a 24-hour blood pressure monitor. Beginning at approximately 7 pm, blood pressure will be measured every 15 minutes. During sleeping hours, blood pressure will be measured every 30 minutes. Subjects will then go home with the blood pressure monitor and will return it to the GCRC that evening at approximately 7 pm.55 In 2005, Schneider et al published a study showing that transcendental meditation decreased levels of hypertension in African Americans with hypertension over a one year time period.9 We, therefore, hypothesize that the nocturnal blood pressure dip will be lower in the treatment group after mindfulness training than in the control group.

   SCREENING LABS

   Thyroid stimulating hormone (TSH):

   Hypothyroidism is a cause of secondary obesity, while hyperthyroidism is a cause of secondary weight loss. While the only exclusionary criteria for this pilot study is a BMI <35, information on participants' thyroid status is important in the ultimate trend analysis of our pilot data.

   Salivary late night cortisol:

   Cushing's syndrome is as an etiology of obesity that alters metabolism and prevents weight loss. Any person with an elevated salivary late night cortisol level will be excluded from the study.

   INPATIENT VISIT PROCEDURES/TIME LINE FOR 24 TOTAL SUBJECTS 1800 hrs Admission 1800 hrs standard meal 1800-2200 hrs blood pressure measurements every 30 minutes 2000 hrs begin overnight fast 2200-0800 hrs blood pressure measurements every 60 minutes 0800-0900 hrs blood pressure measurements every 5 minutes 0800 hrs BIA, H/W ratio, BXA 0830 hrs blood draw 1 (glucose, insulin, cortisol, adiponectin, PAI-1, hsCRP, lipids, IL-6, TNF-alpha) 0835 hrs 75-gram glucola drink 0835-1030 hrs complete psychometric surveys, diet counseling. 1035 hrs blood draw 2 (glucose, insulin, cortisol) 1045 hrs standardized breakfast 1130 hrs discharge

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women between the ages of 55 and 70 without untreated medical illness
* Fluency in the English language
* Body mass index (BMI) ≥30 kg/m2
* Able to walk for at least 10 minutes without needing to stop or without symptom onset

Exclusion Criteria:

* Significant untreated medical illness as evidenced by abnormal electrolytes or liver function tests
* Systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than or equal to 95 mmHg with or without treatment
* Abnormal thyroid stimulating hormone
* Abnormal late night salivary cortisol
* Untreated diabetes mellitus
* Any severe psychiatric condition
* Loss or gain of greater than or equal to 4 pounds in the past 6 months
* Pharmacologic treatment for weight loss within three months before screening
* Treatment with a very low calorie diet within six months before screening
* Use of systemic corticosteroids within three months
* Use of neuroleptic agent within three months
* Treatment for eating disorder within five years
* Diagnosis of a malignant disease except basal cell carcinoma within five years
* Change in smoking status within three months or during course of study
* Any condition that may preclude informed consent

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Decreases in body mass index | Baseline, 6 month, 4 months, 9 months, 1 year

IPD SHARING:
Plan to Share IPD: No